CLINICAL TRIAL: NCT06961292
Title: The Clinical Efficacy of Anterolateral Complex Augmentation in Patients With ACL Rupture Combined With Excessive Internal Tibial Rotation Subluxation: A Bidirectional Cohort Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2024140; M2024141
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: anterior cruciate ligament; anterolateral complex; ateral extra-articular tenodesis; internal rotational tibial subluxation; tibiofemoral position; magnetic resonance imaging; bidirectional cohort study
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Patients who underwent primary anterior cruciate ligament reconstruction at our institution and met the following criteria:
  A. Inclusion Criteria:
  Age ≥ 18 years; Primary unilateral ACL rupture; Preoperative knee MRI completed at our institution; Diagnosis of excessive internal tibial rotation subluxation (EIRTS) based on preoperative MRI measurements (i.e., internal rotation tibial subluxation [IRTS] > 5.8 mm); Patient has been informed of the study details and has provided written informed consent to participate in this cohort study.
  B. Exclusion Criteria:
  Concomitant injury to the medial collateral ligament (MCL), lateral collateral ligament (LCL), or posterior cruciate ligament (PCL); History of contralateral knee injury; History of patellar dislocation; History of prior knee surgery.
- ALC augmentation group: Patients who underwent anterior cruciate ligament reconstruction combined with anterolateral complex augmentation using lateral extra-articular tenodesis (LET) and met the following criteria: A. Inclusion Criteria: Age ≥ 18 years; Primary unilateral ACL rupture; Preoperative knee MRI completed at our institution; Diagnosis of excessive internal tibial rotation subluxation (EIRTS) based on preoperative MRI measurements (i.e., internal rotation tibial subluxation [IRTS] > 5.8 mm); Patient has been informed of the study details and has provided written informed consent to participate in this cohort study. B. Exclusion Criteria: Concomitant injury to the medial collateral ligament (MCL), lateral collateral ligament (LCL), or posterior cruciate ligament (PCL); History of contralateral knee injury; History of patellar dislocation; History of prior knee surgery.

SUMMARY:
This project aims to establish a high-quality, large-scale, single-center bidirectional cohort study to evaluate the postoperative clinical efficacy of ACLR combined with ALC augmentation in a specific high-risk population-patients with ACL rupture exhibiting excessive internal tibial rotation subluxation (EIRTS) on preoperative MRI. The study population will consist of patients with primary ACL rupture, and high-risk individuals will be identified based on the presence of EIRTS on preoperative knee MRI. The exposure group will undergo ACLR combined with ALC augmentation, while the control group will receive standard ACLR. Observational indicators will include all baseline patient characteristics and postoperative clinical outcomes.

DETAILED DESCRIPTION:
Anterior cruciate ligament (ACL) rupture is one of the most common sports injuries in the field of sports medicine and significantly impairs athletic function. Autologous hamstring tendon single-bundle ACL reconstruction (ACLR) is the standard surgical technique for treating ACL rupture. Although most patients can return to sports postoperatively, a subset still experiences graft re-rupture, residual rotational instability of the knee, and other cases of reconstruction failure. Recent studies suggest that concomitant injury to the anterolateral complex (ALC) of the knee may be an important contributing factor. However, there is currently a lack of clinical evidence regarding the diagnosis of ALC injuries and the surgical indications for their treatment. Therefore, whether ALC should be augmented (diagnostic and surgical indications) in addition to routine ACLR, and how it should be augmented (surgical techniques), has become a key focus of current research.

This project aims to establish a high-quality, large-scale, single-center bidirectional cohort study to evaluate the postoperative clinical efficacy of ACLR combined with ALC augmentation in a specific high-risk population-patients with ACL rupture exhibiting excessive internal tibial rotation subluxation (EIRTS) on preoperative MRI. The study population will consist of patients with primary ACL rupture, and high-risk individuals will be identified based on the presence of EIRTS on preoperative knee MRI. The exposure group will undergo ACLR combined with ALC augmentation, while the control group will receive standard ACLR. Observational indicators will include all baseline patient characteristics and postoperative clinical outcomes.

The study includes two follow-up time points: 2 years and 5 years postoperatively. Follow-up will be conducted via outpatient visits and telephone interviews. Based on the follow-up outcomes, multivariate regression models will be used to analyze the association between exposure and clinical outcomes.

This cohort study aims to address treatment strategies for high-risk ACL rupture patients with preoperative EIRTS, thereby improving perioperative management and clinical decision-making in ACL injuries. It will provide important clinical evidence for establishing surgical indications for ALC augmentation and contribute to the development of long-term clinical prediction models for graft failure after ACLR. The findings will support innovation in ACL reconstruction techniques, optimization of perioperative strategies, reduction in postoperative graft failure rates, and improvement in return-to-sport rates. This study holds significant implications for advancing clinical research in the field of sports medicine.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years; Primary unilateral ACL rupture; Preoperative knee MRI completed at our institution; Diagnosis of excessive internal tibial rotation subluxation (EIRTS) based on preoperative MRI measurements (i.e., internal rotation tibial subluxation [IRTS] > 5.8 mm); Patient has been informed of the study details and has provided written informed consent to participate in this cohort study.

Exclusion Criteria:

* Concomitant injury to the medial collateral ligament (MCL), lateral collateral ligament (LCL), or posterior cruciate ligament (PCL); History of contralateral knee injury; History of patellar dislocation; History of prior knee surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent primary anterior cruciate ligament reconstruction at our institution and fulfilled the predefined inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 335 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Graft Failure Rate | At 2 and 5 years postoperatively
  Graft failure was identified based on physical examination findings and postoperative MRI scans at the designated follow-up time points.
Return to Pivoting Sports: Rate and Time | At 2 and 5 years postoperatively
  The rate and timing of return to pivoting sports were recorded at each follow-up time point.

SECONDARY OUTCOMES:
Patient-Reported Outcome Measures | At 2 and 5 years postoperatively
  Patient-reported outcome measures (PROMs) were collected at each follow-up time point using standardized questionnaires, including the Visual Analogue Scale for Pain (VAS), Tegner Activity Score, modified Lysholm Knee Scoring Scale, and the International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form.
Physical Examinations | At 2 and 5 years postoperatively
  Physical examinations were performed at each follow-up visit, including the anterior drawer test, Lachman test, pivot-shift test, and KT-2000 arthrometer assessment.
Muscle Strength | At 2 and 5 years postoperatively
  Isokinetic muscle strength testing of the knee extensors and flexors was performed using the Biodex system.
MRI Measurements | At 2 and 5 years postoperatively
  Postoperative MRI scans were scheduled for all patients to assess tibiofemoral position, osteoarthritis progression, and ACL graft signal intensity as indicators of graft healing, including anterior tibial subluxation (ATS), internal rotational tibial subluxation (IRTS), cartilage thickness and the signal-to-noise quotient (SNQ).

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No